CLINICAL TRIAL: NCT05622942
Title: Randomized, Blinded, Positive-controlled Phase Ib Clinical Trial for Preliminary Evaluation of Safety and Immunogenicity of Recombinant Pneumococcal Protein Vaccine in Adults Aged 50 Years and Older After Vaccination
Brief Title: Clinical Trial of Recombinant Pneumococcal Protein Vaccine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CanSino Biologics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CTP-PBPV-002
Record Dates: First submitted 2022-11-03; First posted 2022-11-21 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Pneumonia; Respiratory Tract Diseases; Respiratory Tract Infections
Keywords: Vaccine; PspA; Pneumolysin; Safety; Immunogenicity; >=50 years
MeSH Terms: conditions — Pneumonia; Respiratory Tract Diseases; Respiratory Tract Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Recombinant Pneumococcal Protein Vaccine（PBPV） (Experimental): Subjects received 1 dose of PBPV
  Interventions: Biological: PBPV
- Pneumococcal Polysaccharide Vaccine-23-valent (PPV23) (Active Comparator): Subjects received 1 dose of PPV23
  Interventions: Biological: PPV23

INTERVENTIONS:
Biological: PBPV — Intramuscular injection, 1 dose of 0.5ml inoculated on day 0
  Arms: Recombinant Pneumococcal Protein Vaccine（PBPV）
Biological: PPV23 — Intramuscular injection, 1 dose of 0.5ml inoculated on day 0
  Arms: Pneumococcal Polysaccharide Vaccine-23-valent (PPV23)

SUMMARY:
Streptococcus pneumoniae infections often cause serious health problems, especially in infants and the elderly. Failure to cover all polysaccharide types of vaccines is a greater problem for adults than for children.

The purpose of this study was to preliminarily evaluate the safety and immunogenicity of a recombinant pneumococcal protein vaccine applied to adults aged 50 years and older to provide a basis for subsequent clinical trial design.

DETAILED DESCRIPTION:
The risk of Streptococcus pneumoniae infection varies widely with age, underlying disease, and living environment. Worldwide, infants and the elderly are at high risk for pneumococcal disease. Disease from pneumococcal infections can affect multiple organ systems and lead to multiple disease syndromes. This vaccine has a higher coverage rate, capable of reaching more than 94%. With the high coverage rate, it can effectively prevent the occurrence of serotype substitution and the outbreak of antibiotic-resistant pneumococcal-associated diseases.

This clinical trial is a Phase Ib clinical trial in adults aged 50 years and older based on the Phase Ia clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Adults 50 years and older at the time of screening
* Willingness to provide legal proof of identity
* Ability to understand the clinical study and voluntarily sign an informed consent form and complete a 6-month follow-up
* Ability to comply with the requirements of the clinical research protocol

Exclusion Criteria:

* Fever, axillary body temperature >37.0℃ before vaccination
* Positive human immunodeficiency virus (HIV) screening
* History of epilepsy, convulsions or seizures or a history of psychiatric illness or family history
* Received immunosuppressive therapy, cytotoxic therapy, glucocorticoid therapy (excluding topical therapy, surface therapy for acute uncomplicated dermatitis, spray therapy for allergic rhinitis) within the past 6 months (interval <6 months)
* Suffering from serious chronic diseases or conditions in progress that can't be controlled smoothly, such as serious cardiovascular diseases, chronic hemolytic anemia, thyroid diseases, etc. (except thyroid nodules)
* History of severe anaphylactic reactions (e.g., systemic allergic reactions) to any component of the test drug and/or history of serious adverse reactions associated with other vaccines, such as allergy, urticaria, dyspnea, angioneurotic edema, or abdominal pain
* People with hypertension that cannot be controlled by medication (when measured on site: systolic blood pressure ≥ 160 mmHg, diastolic blood pressure is ≥ 100 mmHg)
* Pre-immune hemoglobin, white blood cell count, alanine aminotransferase, aspartate aminotransferase, total bilirubin, creatine phosphokinase (CPK), and troponin (CTN) test results are abnormal and are judged by the investigator to be clinically significant
* Positive urine pregnancy test or lactating women, volunteers or their partners planning to become pregnant
* Diseases caused by Streptococcus pneumoniae such as pneumococcal pneumonia, pneumococcal meningitis, etc. within the last 5 years
* Allergic persons, such as those who are allergic to two or more drugs or foods or those who are severely allergic to one drug or food
* Immunocompromised individuals with known or suspected congenital/acquired immunodeficiency as determined by medical history and/or physical examination, uncontrolled autoimmune diseases, etc
* Abnormal coagulation (e.g., clotting factor deficiency, coagulopathy, platelet abnormalities) or significant bruising or clotting disorders
* No spleen or splenectomy due to any condition
* Acute attack of various acute or chronic diseases within the last 7 days
* Pneumococcal vaccination within the last 5 years
* Received or planned to receive blood/plasma products or immunoglobulins during the study period or 3 months prior to vaccination
* Received or plan to participate in an interventional study, receive another investigational drug, vaccine or treatment during the study within the last 1 month
* Received live attenuated vaccine within the last 14 days
* Received subunit vaccine or inactivated vaccine within the last 7 days
* Those planning to have surgery during the study period
* Subject has any other factors that, in the judgment of the investigator, make them unsuitable for participation in the clinical trial

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-03-11 (Actual); Primary Completion 2023-09-14 (Actual); Study Completion 2024-01-30 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse reactions 0~7 days after vaccination | 0~7 days after vaccination
Incidence of adverse reactions 0~30 days after vaccination | 0~30 days after vaccination
Positive (4-fold change) rate of serum Pneumococcal surface protein A(PspA)-RX1, PspA-3296, PspA-5668 and PlyLD protein antibodies at day 30, 3 months and 6 months after vaccination | Day 30, 3 months and 6 months after vaccination

SECONDARY OUTCOMES:
Incidence of adverse reactions within 30 minutes after vaccination | 30 minutes after vaccination
Incidence of adverse events within 30 days after vaccination | 30 days after vaccination
Incidence of Serious Adverse Event (SAE) within 6 months after vaccination | 6 months after vaccination
Evaluation of the incidence of abnormal laboratory hematology values, including hemoglobin, white blood cell count, alanine aminotransferase (AT), aspartate AT, total bilirubin, creatine phosphokinase , before and on day 8 of the subject's exemption | Before and on day 8 of the subject's exemption
Serum PspA-RX1, PspA-3296, PspA-5668, PlyLD protein antibody Geometric Mean Titer (GMT) at 30 days, 3 months and 6 months before and after vaccination | 30 days, 3 months and 6 months before and after vaccination
Serum PspA-RX1, PspA-3296, PspA-5668, PlyLD protein antibody Geometric Mean Increase (GMI) at 30 days, 3 months and 6 months before and after vaccination | 30 days, 3 months and 6 months before and after vaccination
Serum Ply antibody neutralization test activity at 30 days, 3 months and 6 months before and after vaccination | 30 days, 3 months and 6 months before and after vaccination
GMT of serotype specific Multiplexed Opsonophagocytic Killing Assay (MOPA) at 30 days, 3 months and 6 months before and after vaccination | 30 days, 3 months and 6 months before and after vaccination
Positive conversion rate of serotype specific Multiplexed Opsonophagocytic Killing Assay (MOPA) at 30 days, 3 months and 6 months before and after vaccination | 30 days, 3 months and 6 months before and after vaccination
GMI of serotype specific Multiplexed Opsonophagocytic Killing Assay (MOPA) at 30 days, 3 months and 6 months before and after vaccination | 30 days, 3 months and 6 months before and after vaccination

CONTACTS AND LOCATIONS:
Locations (1):
- Lancang Lahu Autonomous County Center for Disease Control and Prevention, Puer, Yunnan, China

IPD SHARING:
Plan to Share IPD: No
In order to maintain the rights of the subject, do not open the Individual Participant Data (IPD)